CLINICAL TRIAL: NCT02587585
Title: An International Randomized Clinical Trial of Activity Feedback During In-patient Stroke Rehabilitation Enabled by Smart Watches
Brief Title: The Effect of Activity Feedback Enabled by Smart Watches During In-patient Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Collaborators: Oxford Brookes University (Other); Oxford International Rehabilitation Foundation and Innovation (Unknown); University of Warwick (Other)
Responsible Party: Principal Investigator, Dr Derick Wade, Professor in Neurological Rehabilitation, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChiECRCT-20150034
Record Dates: First submitted 2015-09-30; First posted 2015-10-27 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomised, parallel group, single-blinded, attention and feedback controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients wear identical watches; one gives no feedback on activity levels and one gives feedback on a two-hourly basis, with progress against a target derived from activity 24 hours earlier.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback against tailored target (Experimental): For each two hour epoch, the watch calculate the level of activity for the same epoch the day before, and adds 5% as the new target to be achieved.
  Interventions: Behavioral: Feedback against tailored target
- No Feedback (Sham Comparator): For participants assigned to the control group, the smart watch will not provide any activity feedback against a target; it simply shows which two hour epoch a person is in.
  Interventions: Behavioral: No feedback

INTERVENTIONS:
Behavioral: Feedback against tailored target — Participants will wear a smart watch every weekday for nine hours during in-patient rehabilitation to monitor activity levels while receiving their usual care. In the active group, the watch will summate activity movement in two hour epochs and the target for the day for that epoch is the activity in the same epoch 24 hours earlier, plus 5%. During an epoch the patient is shown progress towards the target at at the end of an epoch, they will see their final process towards target for that epoch.
  Arms: Feedback against tailored target
Behavioral: No feedback — Participants will wear a smart watch every weekday for nine hours during in-patient rehabilitation to monitor activity levels while receiving their usual care. However the watch face will simply show which epoch a person is in. The watch will collect the activity in exactly the same way over the day.
  Arms: No Feedback

SUMMARY:
The amount of activity completed by individuals within rehabilitation programs, even when units are well staffed, is often far below that required for optimal stroke rehabilitation, and is not individually adapted on a day-to-day basis. Daily feedback on their activity levels may motivate stroke survivors to engage in greater skills practice and thus outcome after stroke. To date only a few trials suggests that augmented feedback may be effective. There is a need for a large pragmatic trial to explore the impact of augmented activity feedback on top of their standard care. The purpose of this study is to determine the effect of augmented activity feedback by smart watches to support in-patient stroke rehabilitation.

DETAILED DESCRIPTION:
This study had a feasibility and pilot development phase from September 2015 to April 2016, and then moved into the main study with some changes in design and execution occurring in the light of experience. Its execution has also been constrained by external factors beyond control.

It is in essence asking whether wearing a Smart Watch which gives feedback on activity every two hours, with a specific target tailored to the patient's performance 24 hours earlier will be associated with a higher rate of physical activity than seen in people wearing the same watch without and feedback been given.

The intervention only lasts unto 21 days, but earlier discharge will terminate that patient's participation sooner. A telephone interview at 12 weeks after entry collect data on mobility.

Outcome measures will assess mobility, activity, and health status.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute/sub-acute in-patient neurorehabilitation of a first stroke at the 2nd affiliated hospital of Anhui University of Traditional Medicine and Acupuncture, Hefei, China.
* Time from onset of stroke to admission for rehabilitation <16 weeks.
* Ability to follow a two stage command; pick up an object, put object on table.
* Independent in mobility prior to admission. Subjects can use any type of assistive device and brace needed.
* Able to understand and repeat information related to the Informed Consent.

Exclusion Criteria:

* Admission for second stroke.
* Subjects who are unable to provide consent due to a cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in activity counts as measured by a triaxial accelerometer from a smart watch from admission to 3 weeks or discharge from rehabilitation | Baseline, Three weeks or at discharge from in-patient rehabilitation if sooner

SECONDARY OUTCOMES:
Activity goal attainment as measured and provided by the smart watch | At three weeks, or discharge if sooner
  Participants in feedback group receive a preset activity goal based on their previous activity levels at baseline. The smart watch will then provide graduated encouragement by increasing their activity goal by about 5%. Every 10-15 minutes the screen lights up and participants can see their activity progress expressed by activity bars (representing 0-100%). Participants reaching their activity goal is used to measure goal attainment.
Change in walking mobility | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner
  Change in walking speed and spatio-temporal characteristics of walking as measured by an inertial sensor on the lower trunk during a 10m walk test.
Fatigue | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner
  Fatigue Severity Index
Health status on EQ-5D-5L | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner, and 12 weeks (by telephone)
  This scale is used a measure for health status and compromises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Change in functional mobility as measured by Rivermead Mobility Index (RMI) | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner, and 12 weeks (by telephone)
  This scale assesses functional mobility in gait, balance and transfers after stroke
Change in cognitive function as measured by The Montreal Cognitive Assessment (MoCA) | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner
  This is a screening instrument for to measure mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Change in arm function recovery | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner
  Grip dynamometer
Change in performance of activities of daily living as measured by Barthel ADL Index | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner
  This scale is used to record what the participant undertakes in personal activities, to establish a degree of independence from any help, physical or verbal.
Change in disability as measured by WHO Disability Assessment Scale (12 item version) | Baseline, Three weeks or discharge from in-patient rehabilitation if sooner, and 12 weeks
  This scale provides a global measure of disability covering 6 domains: cognition, mobility, self-care, getting along, life activities, and participation
Adverse events | At three weeks, or discharge if sooner and at 12 weeks
  Self-reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Derick T Wade, MD, Principal Investigator — Oxford Brookes University
Locations (1):
- The 2nd Affiliated Hospital to Anhui University of Tranditional Chinese Medicine, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided
In the unlikely event that someone asks, it will probably be shared but so far (March 2017) there is no plan

REFERENCES:
- [Derived] Lawrie S, Dong Y, Steins D, Xia Z, Esser P, Sun S, Li F, Amor JD, James C, Izadi H, Cao Y, Wade D, Mayo N, Dawes H; Smart Watch Activity Feedback Trial Committee (SWAFT). Evaluation of a smartwatch-based intervention providing feedback of daily activity within a research-naive stroke ward: a pilot randomised controlled trial. Pilot Feasibility Stud. 2018 Oct 6;4:157. doi: 10.1186/s40814-018-0345-x. eCollection 2018. PMID 30323946
- [Derived] Dong Y, Steins D, Sun S, Li F, Amor JD, James CJ, Xia Z, Dawes H, Izadi H, Cao Y, Wade DT; Smart watch activity feedback trial committee (SWAFT). Does feedback on daily activity level from a Smart watch during inpatient stroke rehabilitation increase physical activity levels? Study protocol for a randomized controlled trial. Trials. 2018 Mar 9;19(1):177. doi: 10.1186/s13063-018-2476-z. PMID 29523170